CLINICAL TRIAL: NCT03738280
Title: Role of EUS in Differential Diagnosis and Malignancy Prediction of Non-hypovascular Solid Pancreatic Lesions: A Prospective Observational Study
Brief Title: Non-hypovascular Solid Pancreatic Lesions: Role of EUS
Acronym: LE-VASC
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Stefano Francesco Crinò, MD, Principal Investigator, Azienda Ospedaliera Universitaria Integrata Verona
Other Study IDs: 1296CESC
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Solid Pancreatic Neoplasms; Endoscopic Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Endoscopic ultrasound-fine needle biopsy — Patients with non-hypovascular solid pancreatic lesion undergo endoscopic ultrasound-fine needle biopsy

SUMMARY:
Vascular pattern of solid pancreatic lesions (SPLs) has been investigated by different abdominal imaging modalities and by contrast-enhanced endoscopic ultrasonography (CE-EUS). Compared with surrounding pancreatic parenchyma three different patterns have been described: hypo-, iso-, and hypervascular. The majority of SPLs are hypovascular, and the diagnostic relevance of hypoenhanced pattern to predict pancreatic adenocarcinoma (PDAC) is well established. Differently, iso- and hypervascular pattern is not specific and can be expressed by several SPLs, with different clinical behavior and management. To date, poor is know about the role of EUS in differential diagnosis of non-hypovascular SPLs and features associated with malignancy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of one or more solid pancreatic lesions preliminary evaluated by contrast-enhanced computed tomography (CE-CT) and/or contrast enhanced magnetic resonance imaging (CE-MRI) reporting a non-hypovascular contrast pattern (e.g., iso- or hypervascular).

Exclusion Criteria:

* Patients with associated chronic pancreatitis features (e.g., pancreatic calcifications)
* Lesion with hypovascular pattern at CE-EUS.
* Lesion not found or non pancreatic at EUS.
* Patients refusing to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients fulfilling inclusion and exclusion criteria will be included in the study.
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Upstream dilation of the main pancreatic duct | 6 months
  Percentage of cases with upstream dilation of main pancreatic duct will be recorded.
Vascular pattern (iso or hypervascular) | 6 months
  Percentage of cases with iso-vascular or hyper-vascular pattern will be recorded.
Lesion borders (smooth or irregular) | 6 months
  Percentage of cases with smooth or irregular borders will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Stefano Francesco Crinò, Verona, VR, Italy

IPD SHARING:
Plan to Share IPD: No